CLINICAL TRIAL: NCT00665015
Title: Pleural Effusions Following Cardiac Surgery: Prevalence, Risk Factors and Clinical Features.
Brief Title: Pleural Effusion Following Cardiac Surgery: Prevalence, Risk Factors and Clinical Features
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Louis-Philippe Boulet, Respirologist, Unité de Recherche en Pneumologie, Hôpital Laval
Other Study IDs: PEFCS-summer 07
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2008-04-23 (Estimated); Status verified 2008-04

CONDITIONS: Pleural Effusion; Coronary Artery Bypass
Keywords: pleural effusion; coronary artery bypass; heart valve replacement
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Pleural effusion is a common complication of cardiac surgery. The aim of this study was to determine the prevalence, characteristics and determinants of clinically significant pleural effusions, defined as those requiring therapeutic pleural drainage.

DETAILED DESCRIPTION:
This was a retrospective cohort study of prevalence and characteristics of patients who had a pleural effusion after coronary artery bypass graft, valve replacement or both procedures.

Information was collected on all consecutive patients who underwent CABG surgery and/or valve replacement between January 1, 2004 and December 31, 2005. Demographic information, anthropometric parameters, cardiac and renal function assessments, and comorbid conditions were retrieved from medical files. We also collected data on the type of procedure, whether it was elective or urgent, the number and origin of the grafts, the duration of surgery and of cardiopulmonary bypass and the postoperative complications, including pleural effusions. Clinical presentation and evolution of the effusions as well as pleural fluid characteristics were also studied.

Patients were considered to have a clinically significant pleural effusion when they met at least one of the following criteria: need for thoracentesis, a pleural drainage tube or a hospital readmission due to a pleural effusion that occurred within one year of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery bypass grafting (CABG)
* Valve replacement
* Combined CABG and valve replacement
* between January 1st, 2004 and December 31st, 2005

Exclusion Criteria:

* Previous CABG
* Pulmonary and/or aortic artery surgery
* Heart or lung transplant
* Pleural effusion present at the time of surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing coronary artery bypass grafting surgery, heart valve replacement surgery or both procedures.
Sampling Method: Non-Probability Sample
Enrollment: 2892 (Actual)
Dates: Start 2004-01; Primary Completion 2005-12 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Pleural effusion requiring therapeutic drainage | within the first 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Philippe Boulet, MD, FRCP(C), Principal Investigator — Unité de Recherche en Pneumologie, Hôpital Laval
Locations (1):
- Unité de Recherche en Pneumologie, Hôpital Laval, Québec, Quebec, Canada

REFERENCES:
- [Derived] Labidi M, Baillot R, Dionne B, Lacasse Y, Maltais F, Boulet LP. Pleural effusions following cardiac surgery: prevalence, risk factors, and clinical features. Chest. 2009 Dec;136(6):1604-1611. doi: 10.1378/chest.09-0689. Epub 2009 Jul 6. PMID 19581352